CLINICAL TRIAL: NCT05320250
Title: Raman Spectroscopy Analysis of Saliva and Salivary Extracellular Vesicles as New Biomarkers for Parkinson's Disease and Atypical Parkinsonisms.
Brief Title: Saliva and Extracellular Vesicles for Parkinson's Disease
Acronym: RaSPiD
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Azienda Ospedaliero Universitaria di Cagliari (Other)
Responsible Party: Sponsor
Other Study IDs: FDG_Saliva_Parkinson_RaSPiD
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-01

CONDITIONS: Parkinson's Disease and Parkinsonism
Keywords: saliva; Raman spectroscopy; extracellular vesicles; rehabilitation biomarkers; diagnosis
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva containing DNA. DNA will not be analysed separatly
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Parkinson's disease: 60 patients. People with Parkinson's disease (pwPD) will be recruited for the study at Fondazione Don Gnocchi.
  PwPD will be assigned to a rehabilitation program that will last for 6 consecutive weeks. Two possible rehabilitation plans are included:
  1. Rehabilitation treatment at the IRCCS S. Maria Nascente: 30 sessions / 5 days a week including motor rehabilitation, cognitive rehabilitation and speech therapy rehabilitation.
  2. Self-treatment program consisting of stretching and active mobilization exercises at home. Before starting the program, the subjects will undergo an educational and training session with the physiotherapist to learn the correct way of carrying out the proposed exercises.
  Interventions: Other: Saliva collection, longitudinal
- Atypical Parkinsonism: Progressive supranuclear palsy: 20 patients; Corticobasal syndrome: 20 patients; Multisystemic atrophy: 20 patients.
  Interventions: Other: Single saliva collection
- REM sleep Behavior Disorder: 30 patients
  Interventions: Other: Single saliva collection
- Healthy controls: 30 patients
  Interventions: Other: Single saliva collection

INTERVENTIONS:
Other: Single saliva collection — 1 ml of saliva will be collected with Salivette swabs.
  Groups: Atypical Parkinsonism; Healthy controls; REM sleep Behavior Disorder
Other: Saliva collection, longitudinal — 1 ml of saliva will be collected with Salivette swabs. Subjects diagnosed with PD will undergo assessments and saliva sampling before starting rehabilitation treatment (T0), at the end of treatment (T1) and 3 months after the end of treatment (T2).
  Groups: Parkinson's disease

SUMMARY:
Rehabilitation is crucial in the treatment of people with Parkinson's disease (PD) as it can ameliorate motor and non-motor impairments, improving their clinical profile and quality of life. Considering the complex biological processes occurring in PD brain, the identification of accessible and measurable biomarkers to monitor the events induced by intensive rehabilitation would help in i)testing rehabilitation effectiveness, ii)improving the design of clinical trials and iii)personalizing the rehabilitation strategies by the prediction of patients' responsiveness. The objective of this project is the validation of Raman analysis of saliva and salivary extracellular vesicles (EV) for the differential diagnosis of Parkinson's disease (PD) and atypical Parkinsonism. The proposed diagnostic method can be integrated in the preliminary assessment and monitoring of the patient by providing a quickly and repeatable measurable biomarker. In the end, this will bring tothe personalization of the rehabilitation path and provide an indication on the outcome of the rehabilitation treatment.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder characterized by motor symptoms such as bradykinesia, tremor, rigidity and postural instability. An accurate rehabilitation program designed considering the specific characteristics of the patient allows you to maximize the effect of drug therapy, improve the patient's quality of life, while also limiting secondary complications related to the progression of the disease. At the time of diagnosis, however, it is particularly important to be able to quickly identify individuals with idiopathic Parkinson's and distinguish them from those who have an atypical form of Parkinsonism, such as Progressive Supranuclear Palsy (PSP), Multiple System Atrophy (MSA), Corticobasal Degeneration (CBD) and Dementia with Lewy bodies (DLB). Atypical Parkinsonisms are in fact progressive diseases that share some signs and symptoms with PD, however these patients do not respond as effectively to drug therapy since the cellular and degenerative mechanisms that characterize them are very different. For these reasons, their early identification is particularly important to identify the best pharmacological and rehabilitative path for each patient.

To ensure a more accurate patient profiling that takes into account the individual complex clinical picture, the discovery of a biomarker that can be periodically measured in an easily accessible biofluid would allow for better patient stratification, monitoring of the course of the disease and careful study of the effects of the pharmacological and rehabilitation program as well as its personalization, with a view to precision medicine designed, defined and built on the patient.

The Laboratory of Nanomedicine and Clinical Biophotonics (LABION) of Fondazione Don Gnocchi has been working for years on using innovative methods such as Raman spectroscopy to identify biomarkers of neurodegenerative diseases in easily accessible biological fluids, such as blood and saliva. Raman Spectroscopy (RS) allows to obtain a specific and complete characterization of a specific fluid in a rapid, sensitive and non-destructive way, without particular procedures for the preparation of the sample to be analyzed. In RS the entire spectrum obtained from the sample is used as a highly specific "fingerprint" for the selected sample (eg saliva, blood, serum, cerebrospinal fluid) which represents the diagnostic biomarker. The Raman analysis of saliva has already demonstrated the possibility of profiling patients with progressive pathologies with good accuracy and, specifically, of distinguishing subjects suffering from amyotrophic lateral sclerosis compared to subjects with other types of neurodegenerative diseases.

At the same time, LABION has verified the possibility of characterizing by Raman spectroscopy, the extracellular vesicles (EV) circulating in the blood of patients with PD. Since 2017, LABION has been working on the biochemical study of circulating EVs in the serum of PD patients by analyzing the EVs in spectroscopy and the ability of RS to identify a specific biochemical profile of blood vesicles that correlates with clinical scales has been demonstrated. UPDRS III and Hoehn and Yahr. The analysis of the EVs present in the saliva of patients with PD could help to understand the origin of biochemical alterations in the saliva as well as identify even more specific markers.

Raman spectroscopy is therefore proposed as a useful method for the rapid and comprehensive biochemical characterization of saliva and the vesicular component present within it, without the use of staining and labeling procedures.

The objective of this project is the validation of a specific Raman molecular signature for the different experimental groups, which can lead to the determination of a biomarker useful for the differential diagnosis of people with PD compared to subjects with atypical Parkinsonism, through the analysis of a biological fluid that is not invasive, thus filling the current lack of a measurable biomarker for rapid differential diagnosis and for monitoring the evolution of the diseases.

The rapid identification and differential diagnosis of subjects with Parkinson's disease and atypical parkinsonisms will allow to promptly identify the optimal pharmacological and rehabilitative therapy for each subject, leading to a significant improvement in the quality of life for the patient and, in the future, an increased probability slowing the progression of the disease.

SAMPLE COLLECTION: Saliva collection from all the selected subjects will be performed following the Salivette (SARSTEDT) manufacturer's instructions. Saliva will be obtained from all subjects after an appropriate lag time from feeding and teeth brushing. Pre-analytical parameters (i.e. storage temperature and time between collection and processing), dietary and smoking habit will be properly recorded. Briefly, the swab will be placed in the mouth and chewed for 60 seconds to stimulate salivation. Then the swab will be centrifuged for 2 minutes at 1,000 g to remove cells fragments and food debris. Collected samples will be stored at -80° C.

SAMPLE PROCESSING: For the Raman analysis, a drop of each sample will be casted on an aluminium foil in order to achieve the Surface Enhanced Raman Scattering (SERS).

EV ISOLATION: different isolation methods will be tested for effective EV isolation. Purified EVs will be then concentrated and analysed by means of standard techniques and by Raman spectroscopy following a previously optimized protocol for blood EVs. The experimetal settings will be adapted to the salivary EVs, considering variations in substrate, acquisition time, etc.

DATA COLLECTION: Salivary and EV spectra will be acquired using an Aramis Raman microscope (Horiba Jobin-Yvon, France) equipped with a laser light source operating at 785 nm and 532 nm. The instrument will be calibrated before each analysis using the reference band of silicon at 520.7 cm-1. Raman spectra will be acquired in the region between 400 and 1600 cm-1 for saliva, 500-1800 nad 2600-3200 cm-1 for EVs using a 50x objective. The software package LabSpec 6 (Horiba Jobin-Yvon, France) will be used for the acquisition of spectra.

DATA PROCESSING: All the acquired spectra will be baseline corrected and normalized by unit vector using the dedicated software LabSpec 6. The contribution of the substrate will be removed from each spectra, if necessary. The statistical analysis to validate the method, will be performed using a multivariate analysis approach. Principal Component analysis (PCA) will be performed in order to reduce data dimensions and to evidence major trends. The first 20 resultant Principal Components (PCs) will be used in a classification model, Linear Discriminant Analysis (LDA), to discriminate the data maximizing the variance between the selected groups. The smallest number of PCs will be selected to prevent data overfitting. Leave-one-out cross-validation and confusion matrix test will be used to evaluate the method sensitivity, precision and accuracy of the LDA model. Mann-Whitney will be performed on PCs scores to verify the differences statistically relevant between the analysed groups. Correlation and partial correlation analysis will be performed using the Spearman's test, assuming as valid correlation only the coefficients with a p-value lower than 0.05. The statistical analysis will be performed using Origin2018 (OriginLab, USA).

ROC Curve will be calculated to assess thediagnostic potential of the method.

ELIGIBILITY:
Inclusion Criteria:

For Pakinson's disease: diagnosis following "MDS clinical diagnostic criteria for Parkinson's disease" (Postuma et al. Movement Disorders vol. 30 1591-1601, 2015), with Hoehn&Yahr between 1 and 3.

The diagnosis of Progressive Supranuclear Palsy will be made according to the criteria of the Movement Disorders Society (Höglinger et al. Mov. Disord. 32, 853-864, 2017). The diagnosis of Corticobasal Syndrome will be made according to the 2013 Armstrong criteria (Armstrong et al. Neurology 80, 496-503, 2013).

The diagnosis of multiple system atrophy will be made according to the Gilman criteria of The diagnosis of Behavior Disorder in REM phase will be made according to the criteria of the "International Classification of Sleep Disorders, Third Edition (ICSD-3)".

Exclusion Criteria:

For all the experimental groups considered and for healthy controls, subjects with concomitant chronic and / or inflammatory diseases of the oral cavity, other systemic diseases (eg anemia, cardiovascular or respiratory diseases), oncological or infectious diseases will be excluded.

Vascular parkinsonisms, monogenic parkinsonisms will also be excluded as well as iatrogenic parkinsonisms, parkinsonisms secondary to exposure to known neurotoxins; parkinsonisms secondary to tumor lesions; parkinsonisms due to normotensive hydrocephalus; subjects with a form of dementia, severe speech disorders and other psychiatric and / or neurological pathologies.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PD patients and people with atypical Parkinsonism will be recrutied at the Neurology Rehabilitation Unit of IRCCS S. Maria Nascente of Fondazione Don Gnocchi, before and after the rehabilitation treatment, at IRCCS Don Gnocchi (Florence) and Centro "S. Maria ai Servi" (Parma).
  Subjects with RBD will be recruited at the University of Cagliari - Neurology Complex Operating Unit - Sleep Center.
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Salivary Raman fingerprint of PD and atypical parkinsonism | 15/12/2021 - 30/11/2024
  Differences in the Raman spectra of saliva. Raman spectroscopy analysis of the saliva of patients with PD and atypical Parkinsonisms for the validation of the diagnostic power of the method

SECONDARY OUTCOMES:
Salivary Raman fingerprint of PD patients after rehabilitation | 15/12/2021 - 30/11/2024
  Changes in the Raman spectra of saliva before and after rehabilitation. Raman spectroscopy analysis of the saliva of patients with PD and atypical Parkinsonisms for the validation of the diagnostic power of the method
Salivary Extracellular vesicles characterization | 01/03/2022 - 30/11/2024
  Differences in the Raman spectra of salivary EVs. Isolation and characterization with standard techniques and by Raman spectroscopy of salivary extracellular vesicles
Correlation of Raman data with clinical assessments | 01/10/2022 - 31/12/2024
  Correlation between spectral differences and changes before and after rehabilitation and clinical assessment by Hoehn and Yahr and UPDRS III . Data analysis, correlation study and data interpretation

CONTACTS AND LOCATIONS:
Overall Officials: Alice Gualerzi, PhD, Principal Investigator — Fondazione Don Carlo Gnocchi
Locations (4):
- Italy (4):
  - Azienda Ospedaliero - Universitaria di Cagliari, Cagliari
  - IRCCS Fondazione Don Carlo Gnocchi, Florence
  - IRCCS S. Maria Nascente, Fondazione Don Carlo Gnocchi ONLUS, Milan
  - Fondazione Don Gnocchi, Centro "S. Maria ai Servi", Parma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carlomagno C, Bertazioli D, Gualerzi A, Picciolini S, Andrico M, Roda F, Meloni M, Banfi PI, Verde F, Ticozzi N, Silani V, Messina E, Bedoni M. Identification of the Raman Salivary Fingerprint of Parkinson's Disease Through the Spectroscopic- Computational Combinatory Approach. Front Neurosci. 2021 Oct 26;15:704963. doi: 10.3389/fnins.2021.704963. eCollection 2021. PMID 34764849
- [Background] Gualerzi A, Picciolini S, Carlomagno C, Terenzi F, Ramat S, Sorbi S, Bedoni M. Raman profiling of circulating extracellular vesicles for the stratification of Parkinson's patients. Nanomedicine. 2019 Nov;22:102097. doi: 10.1016/j.nano.2019.102097. Epub 2019 Oct 21. PMID 31648040